CLINICAL TRIAL: NCT01407406
Title: A Single-Dose, Randomized, Double-Blind, Parallel-Group, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BIIB023 in Chinese, Japanese, and Caucasian Adult Healthy Volunteers
Brief Title: Phase 1 Study to Evaluate the PK, Safety, Tolerability of BIIB023 in Chinese, Japanese, and Caucasian Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 211HV102
Record Dates: First submitted 2011-07-14; First posted 2011-08-02 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — BIIB023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Chinese Subjects - low dose BIIB023 IV (Experimental)
  Interventions: Drug: BIIB023 - low dose IV Dose
- Chinese Subjects - high dose BIIB023 IV (Experimental)
  Interventions: Drug: BIIB023 - high dose IV Dose
- Japanese Subjects - low dose BIIB023 IV (Experimental)
  Interventions: Drug: BIIB023 - low dose IV Dose
- Japanese Subjects - high dose BIIB023 IV (Experimental)
  Interventions: Drug: BIIB023 - high dose IV Dose
- Causasian Subjects - low dose BIIB023 IV (Experimental)
  Interventions: Drug: BIIB023 - low dose IV Dose
- Caucasian Subjects - high dose BIIB023 IV (Experimental)
  Interventions: Drug: BIIB023 - high dose IV Dose

INTERVENTIONS:
Drug: BIIB023 - low dose IV Dose
  Arms: Causasian Subjects - low dose BIIB023 IV; Chinese Subjects - low dose BIIB023 IV; Japanese Subjects - low dose BIIB023 IV
Drug: BIIB023 - high dose IV Dose
  Arms: Caucasian Subjects - high dose BIIB023 IV; Chinese Subjects - high dose BIIB023 IV; Japanese Subjects - high dose BIIB023 IV

SUMMARY:
Rationale for the Study: Phase 1 pharmacokinetic (PK) data is needed in Chinese and Japanese populations to support future clinical development of BIIB023 in China and Japan.

Study Design: This is a single-dose study to assess the PK, safety, and tolerability of BIIB023 administered intravenously (IV) to adult Chinese, Japanese, and Caucasian healthy volunteers. The Caucasian group is included to allow comparison of PK data from different groups using data from the same study under the same controlled conditions.

Subjects will be in the clinic for 48 hours around the time of dosing and in the study for up to 100 days.

DETAILED DESCRIPTION:
Rationale for the Study: Phase 1 pharmacokinetic (PK) data is needed in Chinese and Japanese populations to support future clinical development of BIIB023 in China and Japan.

Study Design: This is a single-dose, Randomized, Double-Blind, parallel-group study to evaluate the PK, safety, and tolerability of BIIB023 administered intravenously (IV) to adult Chinese, Japanese, and Caucasian healthy volunteers. The Caucasian group is included to allow comparison of PK data from different groups using data from the same study under the same controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must have the ability to understand the purpose and risks of the study & provide signed & dated informed consent.
* Chinese, Japanese or Caucasian subjects
* Subjects of childbearing potential must practice effective contraception during the study and 3 months after their last dose of study treatment.
* Must have a BMI within the range of 18.5 to 25 kg/m2.
* Must be willing to abstain from using tobacco and tobacco-containing products during the in-clinic period.
* Must be willing to limit alcohol intake to no more than 2 units per day throughout the duration of the study (with some stricter exceptions at various timepoints).
* Must be deemed healthy as determined by the Investigator, based on assessments at Screening and Day -1.

Exclusion Criteria:

* Known to have a positive test result for Human Immunodeficiency Virus (HIV) antibody.
* Known history of hepatitis C or hepatitis B virus.
* History of tuberculosis (TB) or a positive QuantiFERON®-TB Gold test.
* Subjects with a history of carcinoma in situ and malignant disease. (with the exception of basal cell carcinoma that has been completely excised prior to study)
* History of clinically important severe allergic or anaphylactic reactions.
* Known allergy to components of the BIIB023 formulation.
* History of any clinically important cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
* Abnormal hematology or blood chemistry values at Screening or Day -1, as determined by the Investigator.
* Serious infection (e.g., pneumonia, septicemia) within the 2 months prior to Screening.
* History of drug or alcohol abuse (as defined by the Investigator) within 6 months prior to screening, and/or a positive urine drug screen (without a medically indicated rationale) or positive alcohol breath test at Screening or on Day -1.
* Active bacterial or viral infection and fever >38°C within 48 hours prior to study treatment administration.
* Female subjects who are pregnant, currently breastfeeding, or attempting to conceive during the study.
* Surgery within 3 months prior to Day -1 or any surgical procedure planned during the course of the study
* Previous exposure to BIIB023.
* Treatment with another investigational drug , device, or approved therapy for investigational use within 30 days prior to Day -1, or 7 half lives of the investigational product, whichever is longer
* Treatment with any prescription medication within 2 weeks before Day -1 with the exception of oral contraceptives for women of childbearing potential.
* Treatment with any nonprescription medicinal products (including vitamin/mineral/herbal containing preparations but excluding acetaminophen) within the 7 days prior to study treatment.
* Vaccination within 4 weeks of study treatment.
* Blood donation (1 unit or more) within 1 month prior to study treatment or plasma donation within 7 days prior to study treatment.
* Alcohol use within 48 hours prior to study treatment or during the In-Clinic period.
* Current enrollment in any other study treatment or disease study.
* Inability to comply with study requirements.
* Vigorous exercise (as determined by the Investigator) within 72 hours prior to any study visit.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen Idec, make the subject unsuitable for enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
AUC of BIIB023 | Participants will be followed for the duration of a study; an expected 71 days
Cmax of BIIB023 | Participants will be followed for the duration of a study; an expected 71 days
Tmax of BIIIB023 | Participants will be followed for the duration of a study; an expected 71 days
Half-life of BIIB023 | Participants will be followed for the duration of a study; an expected 71 days
Volume of distribution of BIIB023 | Participants will be followed for the duration of a study; an expected 71 days
Clearance of BIIB023 | Participants will be followed for the duration of a study; an expected 71 days

SECONDARY OUTCOMES:
Number of patients with Adverse Events as a measure of safety and tolerability | Participants will be followed for the duration of a study; an expected 71 days
Number of patients with Serious Adverse Events as a measure of safety and tolerability | Participants will be followed for the duration of a study; an expected 71 days

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Melbourne, Victoria, Australia
- Research Site, Hong Kong, Hong Kong, China